CLINICAL TRIAL: NCT01295034
Title: Vitamin D Supplements for HIV-positive Patients on cART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Branch (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Andrea Branch, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 10-0679; R01DA031095 (NIH)
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: HIV-associated Co-morbidities
Keywords: HIV; combination antiretroviral therapy; vitamin D; low bone density
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional vitamin D treatment (Placebo Comparator): Subjects in Protocol A (the conventional/active placebo arm) will receive 50,000 IU/wk of vitamin D2 for 8 wk followed by 1000 IU/d of vitamin D3 for 48 wk.
  Interventions: Dietary Supplement: conventional vitamin D treatment
- tiered/titrated vitamin D dosing (Experimental): Subjects in Protocol B will receive 2000-4000 IU/d of vitamin D3, depending on the basal 25(OH)D level, with dose titration, as necessary, based on the slope of the initial response, for a total duration of treatment of 12 mo.
  Interventions: Drug: tiered/titrated vitamin D dosing

INTERVENTIONS:
Dietary Supplement: conventional vitamin D treatment — Subjects in Protocol A (the conventional/active placebo arm) will receive 50,000 IU/wk of vitamin D2 for 8 wk followed by 1000 IU/d of vitamin D3 for 48 wk.
  Arms: conventional vitamin D treatment
Drug: tiered/titrated vitamin D dosing — Subjects in Protocol B will receive 2000-4000 IU/d of vitamin D3, depending on the basal 25(OH)D level, with dose titration, as necessary, based on the slope of the initial response, for a total duration of treatment of 12 mo.
  Arms: tiered/titrated vitamin D dosing

SUMMARY:
The ability of vitamin D to modulate the immune system and strengthen bones may mitigate the adverse medication consequences of HIV/AIDS, but little is known about either the health benefits of vitamin D supplements, or about the optimal dosing regimen for patients on highly active antiretroviral therapy (HAART). This trial is a comparison of two regimens for administering vitamin D and calcium to HIV-positive individuals taking antiviral medications. This study will help physicians make evidence-based decisions about the most effective way to use vitamin D in their patients and enable the design of large multi-center trials in the future.

DETAILED DESCRIPTION:
In the post-HAART era, patients continue to suffer from the adverse medical consequences of HIV/AIDS. The adverse effects include incomplete immune reconstitution, chronic inflammation, depression, increased risk of cardiovascular and metabolic disease, and low bone density. Clinical trials suggest that vitamin D supplements can increase bone density, reduce inflammation, alleviate depression, and increase longevity if given in adequate doses. To achieve maximum benefits, most vitamin D experts in the HIV field agree that vitamin D treatments should raise the concentration of 25-hydroxyvitamin D [25(OH)D] above 30 ng/ml. A growing number of HIV care providers desire an evidence-based protocol for achieving these 25(OH)D target levels. This project addresses the need for a validated protocol for treating vitamin D deficiency in HIV-positive individuals on HAART. The goal of Aim I is to conduct a 12-mo randomized, double-blinded trial comparing two dosing regimens of oral vitamin D plus 0.5 g/d of calcium in patients on stable HAART who have 25(OH)D levels ≤ 25 ng/ml and undetectable HIV viral load at baseline (100 per arm). Medication event monitoring system (MEMS) caps will be used to record supplement use and to promote adherence. Subjects in Protocol A will receive 50,000 IU/wk of vitamin D2 for 8 wk followed by 1000 IU/d of vitamin D3 for 48 wk. Subjects in Protocol B will receive 2000-4000 IU/d of vitamin D3, depending on the basal 25(OH)D level, with dose titration, as necessary, based on the slope of the initial response. The primary outcome measure is the difference in the percentage of subjects with 25(OH)D levels in the range of 30-60 ng/ml at 12 mo. The secondary outcome is the slope of the 25(OH)D response curve during various time intervals. The goal of Aim II is to compare the impact of the two protocols on markers of disease. The primary outcome measure is the change in the CD4+T cell count. Secondary outcomes include changes in CD4+ T cell subsets, markers of inflammation, markers of bone and calcium metabolism, self-reported psychological status, viral load, side effects, safety, and adherence. To our knowledge, this trial is the first head-to-head comparison of a regimen that uses a loading dose of vitamin D2 with a regimen that uses a tiered starting dose of vitamin D3. The project will yield a validated protocol for treating vitamin D deficiency in HIV-infected patients on HAART and will provide initial data about the risks and health benefits of vitamin D and calcium supplements. This information is essential for designing definitive multicenter trials in the future.

ELIGIBILITY:
Inclusion Criteria:

* age, 18-70 yr
* HIV-infected
* on a stable HAART regimen for at least 12 mo with an undetectable HIV viral load for 6-mo
* willing to participate
* not receiving vitamin D supplementation in a form other than vitamin D2 or vitamin D3
* not receiving treatment for bone disease
* not receiving medications known to alter bone mineralization
* not suffering from conditions known to affect vitamin D, calcium, and/or phosphate levels (including clinically significant hypocalcemia, primary hyperparathyroidism)
* not experiencing kidney disease based on GFR > 60 min/ml/1.73 m2, 10) 25(OH)D level < 25 ng/ml
* not meeting criteria of the National Osteoporosis Foundation for established bone disease (osteoporosis, osteomalacia) requiring immediate treatment
* not consuming more than 2.0 gm of calcium/day in food and supplements combined outside the trial
* not consuming more than 800IU/day of vitamin D outside the trial
* not suffering from an unstable medical condition likely to preclude participation in a 12 month trial
* able to ingest and absorb food and nutrients
* not pregnant or planning to become pregnant.

Exclusion Criteria:

* No history or evidence of HIV infection
* HIV viral load positive
* outside the age range

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea D Branch, PhD, Principal Investigator — Icahn School of Medicine Mount Sinai
Locations (1):
- Icahn School of Medicine Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McComsey GA, Tebas P, Shane E, Yin MT, Overton ET, Huang JS, Aldrovandi GM, Cardoso SW, Santana JL, Brown TT. Bone disease in HIV infection: a practical review and recommendations for HIV care providers. Clin Infect Dis. 2010 Oct 15;51(8):937-46. doi: 10.1086/656412. PMID 20839968

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Vitamin D Treatment: conventional vitamin D treatment: Subjects in Protocol A (the conventional/active placebo arm) received 50,000 IU/wk of vitamin D2 for 8 wk followed by 1000 IU/d of vitamin D3 for 48 wk.
- Tiered/Titrated Vitamin D Dosing: tiered/titrated vitamin D dosing: Subjects in Protocol B received 2000-4000 IU/d of vitamin D3, depending on the basal 25(OH)D level, with dose titration, as necessary, based on the slope of the initial response, for a total duration of treatment of 12 mo.
Period: Overall Study
Arm/Group | Conventional Vitamin D Treatment | Tiered/Titrated Vitamin D Dosing
Started | 32 | 30
Completed | 27 | 25
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Conventional Vitamin B Dosing: Subjects in Protocol A (the conventional/active placebo arm) will receive 50,000 IU/wk of vitamin D2 for 8 wk followed by 1000 IU/d of vitamin D3 for 48 wk.
- Tiered/Titrated Vitamin B Dosing: tiered/titrated vitamin D dosing: Subjects in Protocol B received 2000-4000 IU/d of vitamin D3, depending on the basal 25(OH)D level, with dose titration, as necessary, based on the slope of the initial response, for a total duration of treatment of 12 mo.
- Total: Total of all reporting groups
Arm/Group | Conventional Vitamin B Dosing | Tiered/Titrated Vitamin B Dosing | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 30 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [39 to 51] | 48 [42 to 52] | 48 [41 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: 25(OH)D Levels
Description: The difference in the percentage of subjects with 25(OH)D levels in the range of 30-60 ng/ml at 12 mo between the two arms.
Time Frame: baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Vitamin D Treatment | Tiered/Titrated Vitamin D Dosing
Number analyzed (Participants) | 32 | 30
Participants | 13 | 20

2. Secondary Outcome: CD4+T Cell Count
Description: The change in the CD4+T cell count between the two arms.
Time Frame: baseline and 12 months
Population: Analysis only for participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: cell/μL
Groups:
- Conventional Vitamin B Dosing: Subjects in Protocol A (the conventional/active placebo arm) received 50,000 IU/wk of vitamin D2 for 8 wk followed by 1000 IU/d of vitamin D3 for 48 wk.
Arm/Group | Conventional Vitamin B Dosing | Tiered/Titrated Vitamin D Dosing
Number analyzed (Participants) | 27 | 23
cell/μL | 26 [-56 to 122] | 40 [-45 to 65]

ADVERSE EVENTS:
Groups:
- Tiered/Titrated Vitamin B Dosing: Subjects in Protocol B received 2000-4000 IU/d of vitamin D3, depending on the basal 25(OH)D level, with dose titration, as necessary, based on the slope of the initial response, for a total duration of treatment of 12 mo.
Arm/Group | Conventional Vitamin B Dosing | Tiered/Titrated Vitamin B Dosing
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No